CLINICAL TRIAL: NCT05129995
Title: The Impact of Passive Heat Treatment on Skeletal Muscle Perfusion Capacity and Post-prandial Muscle Protein Synthesis Rates in Healthy Older Adults
Brief Title: Passive Heat Treatment and Skeletal Muscle Reconditioning Older Adults
Acronym: Sauna
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC 21-072
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: single arm, within subject study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passive heat treatment (Experimental): Infrared sauna bathing
  Interventions: Other: Passive heat treatment

INTERVENTIONS:
Other: Passive heat treatment — Participants will be subjected to an 8-week (3 x pw) passive heat treatment, by means of infrared sauna bathing, intervention.
  Other Names: Sauna bathing

SUMMARY:
Rationale: Aging is accompanied by impairments in the sensitivity of skeletal muscle tissue to respond to the anabolic properties of protein feeding, which is suggested to result in age-related loss in muscle mass. Adequate muscle perfusion capacity is essential for muscle mass maintenance, as it determines the rapid delivery of amino acids, nutrients and growth factors to the muscle fiber, thereby stimulating muscle protein synthesis. However, muscle perfusion capacity declines with increasing age. Hence, improving muscle perfusion may be key to augment the sensitivity of senescent muscle following protein feeding in older adults. Although exercise training is an effective way to improve muscle perfusion capacity, there are a number of patient groups that find exercise training difficult to achieve. Hence, alternative strategies need to be developed to improve muscle perfusion capacity. Passive heat treatment (PHT) has been associated with various health benefits in older adult populations, including improved blood pressure, cardiovascular disease risk, and metabolic health. In addition, PHT has been shown to increase muscle fiber capillarization in healthy young adults. However, whether such an intervention improves muscle perfusion capacity, and enhances the anabolic response of skeletal muscle following food ingestion in older adults is unknown.

Objective: To assess the impact of an 8-week passive heat treatment intervention on skeletal muscle fiber capillarization/perfusion capacity and post-prandial muscle protein synthesis rates in healthy older adults.

Study design: single arm, within subject study design

Study population: 14 healthy older (65-85 y) men and women.

Intervention (if applicable): Participants will be subjected to an 8-week (3 x pw) PHT, by means of infrared sauna bathing, intervention. Before and after the PHT intervention the participants will undergo one test day during which blood pressure, body composition, physical function and muscle strength will be assessed. In addition, before and after the PHT intervention period subjects will be complete a 'whole-meal test day' during which the muscle protein synthesis and perfusion capacity response will be evaluated following the ingestion of a whole food meal. Basal and post-prandial muscle protein synthesis and perfusion capacity will be assessed by a continuous infusion of labelled amino acids combined with contrast-enhanced ultrasound measurements. Blood and muscle samples will be collected in order to assess the muscle protein synthetic response.

Main study parameters/endpoints: The primary outcome will be post-prandial muscle protein synthesis rates following meal ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-85 years
* Body mass index 18.5 - 30 kg/m2
* Healthy
* Having given informed consent

Exclusion Criteria:

* Allergy for one of the food items used
* >5% weight change in the previous 6 months
* Participating in a structured (progressive) exercise program, or in the past 3 months.
* Frequent (more than once per week) user of infrared (or traditional) sauna in the past 3 months
* Smoking
* Diagnosed with cardiovascular disease, kidney failure, rheumatoid arthritis
* Diagnosed musculoskeletal, GI tract, metabolic (e.g. diabetes) or pulmonary (e.g. COPD) disorders
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories (NSAIDs).
* Chronic use of gastric acid suppressing medication and/ or anti-coagulants
* Recent (<1 year) participation in amino acid tracer (L-[ring-13C6]-phenylalanine and L-[3,5-2H2]-tyrosine) studies
* Blood donation in the past 2 months
* Strict Following a vegetarian diet
* Known allergic reaction to ultrasound contrast agent
* Non Dutch speaking

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Post-prandial muscle protein synthesis rates | 4 hours following meal ingestion
  Fractional synthetic rates calculated based on tissue-free, plasma, and protein-bound tracer enrichments using stable isotope methodology

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No